CLINICAL TRIAL: NCT01805648
Title: A Multicenter, Single-Arm, Open Label Study Evaluating the Efficacy and Safety of Maintenance Treatment With Recombinant Human Thrombopoietin in Thrombocytopenic Subjects With Immune Thrombocytopenia
Brief Title: Efficacy and Safety Study of Maintenance Treatment With rhTPO in Thrombocytopenic Subjects With ITP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College (Other)
Collaborators: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Principal Investigator, Yongqiang Zhao, The Director of Hematology Department of Peking Union Medical College Hospital, Peking Union Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPOzyq120725
Record Dates: First submitted 2013-02-22; First posted 2013-03-06 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Thrombocytopenia; Immune Thrombocytopenia; Idiopathic Thrombocytopenic Purpura
Keywords: ITP; rhTPO
MeSH Terms: conditions — Thrombocytopenia; Purpura, Thrombocytopenic, Idiopathic | interventions — Thrombopoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rhTPO (Experimental): Active investigational product
  Interventions: Drug: rhTPO

INTERVENTIONS:
Drug: rhTPO — Subcutaneously dosing of rhTPO is based on screening weight. Subjects will be given rhTPO 300 IU/Kg once daily up to 14 days in the pre-treatment period . When two consecutive platelet counts is above 50×10^9/L, the subjects will be begin to receive maintenance treatment of rhTPO 300 IU/Kg. In the period of maintenance treatment, starting dosing interval of rhTPO is every other day followed by the interval adjustments for keeping platelet counts between 30×10^9/L～100×10^9/L.
  Other Names: Recombinant Human Thrombopoietin; Recombinant Human TPO

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of rhTPO in the maintenance treatment of ITP, to explore the appropriate dosing interval of the maintenance treatment of rhTPO .

DETAILED DESCRIPTION:
The eligible subjects with ITP firstly will receive a pre-treatment of rhTPO 300 IU/Kg once daily up to 14 days. The subjects with two consecutive platelet counts above 50×10^9/L in the pre-treatment period will begin to receive maintenance treatment of rhTPO 300 IU/Kg for 12 weeks. In the period of maintenance treatment, starting dosing interval of rhTPO is every other day followed by the interval adjustments for keeping platelet counts between 30 ×10^9/L～100 ×10^9/L. Subsequently, subjects will stop treatment of rhTPO and be followed up for 4 weeks after maintenance treatment.

Platelet count, bleeding and other symptoms will be evaluated before and after treatment.

Platelet transfusion will be administered to subjects with active bleeding symptoms.

Toxicity will be monitored continuously during the entire study. Safety will be assessed by adverse events and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria for immune thrombocytopenia (idiopathic thrombocytopenic purpura).
* Subject with resistance to or relapse after glucocorticoid in the treatment of ITP, not accepts splenectomy, or subject with ineffective or relapse after surgical splenectomy.
* Two consecutive platelet counts (not in the same day) < 30×10^9/L.
* Subject is willing and able to provide written informed consent.

Exclusion Criteria:

* Pregnancy or breast feeding.
* Having a medical history of thrombosis.
* Significant abnormal cardio-pulmonary function.
* Abnormal liver and kidney function:

  * a serum creatinine concentration≥ 176.8µmol/l (1.5mg/dl);
  * a serum aminotransferase concentration: more than 2.0 times the upper limit of the normal range.
  * a serum bilirubin concentration: more than 2.0 times the upper limit of the normal range.
* Synchronous tumor.
* Cannot adopt adequate contraceptive precautions during the course of the study.
* Any other treatment drugs for ITP are being taken (except the duration of reducing glucocorticoid dosage as ineffective treatment ).
* Any other situation that is not suitable for participating in the trial according to the judgment of the investigator .

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The effective rate of maintenance treatment (the platelet count continued to be over 30 × 10^9/L) | up to 16 weeks per subject

SECONDARY OUTCOMES:
The effective rate of maintenance treatments adopting different frequency of administration | up to 16 weeks per subject
Number of subjects with Adverse Events as a Measure of Safety | up to 18 weeks per subject

CONTACTS AND LOCATIONS:
Overall Officials: Yongqiang Zhao, Dr., Principal Investigator — Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Beijing, China